CLINICAL TRIAL: NCT01450358
Title: Evaluation of Antimicrobial Use and Time of Treatment of Nosocomial Sepsis Comparing Polymerase Chain Reaction (PCR) in Real Time Multiplex to the Conventional Blood Culture for Etiologic Agents Identification. Randomized Clinical Trial.
Brief Title: Evaluation in the Treatment of Nosocomial Sepsis Comparing Polymerase Chain Reaction With Conventional Blood Culture.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto do Coracao (Other Government)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Tania Mara Varejão Strabelli, PhD, Director of Infection Control Unit, Instituto do Coracao
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PCR multiplex
Record Dates: First submitted 2011-10-10; First posted 2011-10-12 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Sepsis; Bacteremia; Fungemia
Keywords: Sepsis; Real time PCR; Blood culture; Bacteremia diagnosis; Fungemia diagnosis
MeSH Terms: conditions — Sepsis; Bacteremia; Fungemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pathogen detection by Multiplex PCR (Active Comparator): Blood samples for cultures and Multiplex PCR will be collected before start the antibiotic therapy in patients with sepsis. Multiplex PCR will be immediately undertaken and its results will be reported to prompt medical researcher (6-12 hours).The medical researcher will change the antibiotic regimen (De-escalation) immediately as a result of Multiplex PCR.
  Interventions: Other: Antibiotic regimen
- Pathogen detection by blood culture (No Intervention): Blood samples for cultures and Multiplex PCR will be collected before start the antibiotic therapy in patients with sepsis. The results of multiplex PCR will be not informed to the medical researcher, being focused care as a result of blood culture (at least after 72 hours).

INTERVENTIONS:
Other: Antibiotic regimen — The medical researcher will change the antibiotic regimen (De-escalation) immediately as a result of Multiplex PCR (6-12 h).
  Arms: Pathogen detection by Multiplex PCR

SUMMARY:
The objective of this study is to evaluate the consumption of antimicrobial therapy in patients comparing a rapid molecular test (PCR in Real-Time Multiplex) with blood cultures to identify the etiological agents of sepsis.

DETAILED DESCRIPTION:
Patients staying more than 48 hours in hospital with clinical suspicion of sepsis could be included in the study. Blood samples for cultures and multiplex PCR will be collected immediately prior to initiation of antibiotic therapy. Patients will be randomly selected into two groups. In Group I, the PCR results will be immediately reported to the medical researcher (6-12 hours), which will change the antimicrobial regimen (De-escalation). In Group II, the Multiplex PCR results will not be informed, being focused care as a result of blood culture (at least after 72 hours). The initial empirical antimicrobial therapy will be the same in both groups, according to the standardization of the institution.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 or more years old
* Patient staying more than 48 hours in hospital
* Patient with clinical suspicion of infection and presenting at leat two of the following criteria:temperature > 38oC or < 36oC, heart rate > 90 beats/minute, respiratory rate > 20 breaths/minute or PaCO2 < 32 mmHg or leukocytosis >12 000/μl or leukopenia <4000/μl or normal white blood cell count with >10% immature forms
* Patient or responsible able to provide informed consent

Exclusion Criteria:

* Patient submitted to cardiovascular surgery in the last fifteen days
* Patient or responsible are not able to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of antimicrobial use in number of days comparing a rapid molecular test (PCR in Real-Time Multiplex) with blood cultures to identify the etiological agents of sepsis. | After fourteen days of antimicrobial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tania MV Strabelli, PhD, Principal Investigator — Instituto do Coracao
Locations (1):
- Instituto do Coracao, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Rodrigues C, Siciliano RF, Filho HC, Charbel CE, de Carvalho Sarahyba da Silva L, Baiardo Redaelli M, de Paula Rosa Passetti AP, Franco MRG, Rossi F, Zeigler R, De Backer D, Franco RA, de Almeida JP, Rizk SI, Fukushima JT, Landoni G, Uip DE, Hajjar LA, Strabelli TMV. The effect of a rapid molecular blood test on the use of antibiotics for nosocomial sepsis: a randomized clinical trial. J Intensive Care. 2019 Jul 22;7:37. doi: 10.1186/s40560-019-0391-3. eCollection 2019. PMID 31367384